CLINICAL TRIAL: NCT00937352
Title: A Phase 3 Extension, Multicenter, Double-Blind, Long-Term Safety and Tolerability Treatment Trial of Bapineuzumab (AAB-001, ELN115727) in Subjects With Alzheimer's Disease Who Participated in Study ELN115727-301 or Study ELN115727-302.
Brief Title: A Long-Term Safety and Tolerability Study in Subjects With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELN115727-351
Record Dates: First submitted 2009-07-07; First posted 2009-07-13 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease
Keywords: Mild to moderate Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bapineuzumab 0.5 mg/kg (Active Comparator): 0.5 mg/kg
  Interventions: Drug: Bapineuzumab
- Bapineuzumab 1.0 mg/kg (Active Comparator): 1.0 mg/kg
  Interventions: Drug: Bapineuzumab

INTERVENTIONS:
Drug: Bapineuzumab — 0.5 mg/kg, administered via IV (in the vein) infusion every 13 weeks for 4 years.
  1.0 mg/kg, administered via IV (in the vein) infusion every 13 weeks for 4 years.

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of Bapineuzumab (AAB-001, ELN115727) in subjects with Alzheimer's disease who participated in study ELN115727-301 or study ELN115727-302.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Must have completed study 301 or study 302; and have completed Visit 15 (Week 78)
* Brain MRI scan to evaluate safety from Study 301 or 302 at Visit 14/Week 71
* Caregiver able to attend all clinic visits with patient

Exclusion Criteria:

* Any new medical contraindication or clinically significant abnormality on physical, neurological, laboratory, vital signs or ECG examination (eg, atrial fibrillation) that precludes continued or initiation of treatment with bapineuzumab or participation in the study
* Screening visit brain MRI scan (MRI from Study 301 or 302 Visit 14/Week 71) indicative of any significant abnormality not approved by the medical monitor prior to enrollment
* Current use of experimental medications for AD (other than bapineuzumab) and all other experimental medications, herbal preparations containing Ginko biloba, and anticoagulants (except the use of aspirin 325mg/day or less, Plavix, and Persantine but not for stroke)

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinically important changes in safety assessment results including vital signs, weight, clinical laboratory tests, electrocardiograms (ECGs), brain magnetic resonance imaging (MRI), physical and neurological examinations, and infusion site assessments. | Varies according to assessment: vital signs and adverse events on ongoing basis; MRI and ECG as required per protocol

SECONDARY OUTCOMES:
To evaluate the efficacy of long term treatment of IV administered bapineuzumab in subjects with AD. | The trial duration is expected to be approximately 4 years. The study will last up to the time of commercial launch of bapineuzumab, or termination of the clinical trials program, whichever comes first

CONTACTS AND LOCATIONS:
Locations (191):
- United States (176):
  - University of Alabama Hospital, Birmingham, Alabama
  - Dedicated Clinical Research, Inc., Goodyear, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Banner Research Institute, Sun City, Arizona
  - University of Arizona College of Medicine, Health Sciences Center, Tucson, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - East Bay Physicians Medical Group, Berkeley, California
  - AVI Clinical Research, Carson, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Pharmacology Research Institute, Encino, California
  - Margolin Brain Institute, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Coordinated Clinical Research, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Collaborative NeuroScience Network, Inc., Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - UCLA Department of Neurology, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Neurology Center, Oceanside, California
  - University of California, Irvine Medical Center, Orange, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Sutter Neuroscience Medical Group, Sacramento, California
  - University of California at Davis, Alzheimer's Disease Research Center, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Mile High Research Center, Denver, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Christiana Care Neurology Specialists, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - JEM Research, LLC, Atlantis, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Quantum Laboratories, Inc., Deerfield Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neurologic Consultants, PA, Fort Lauderdale, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Clinical Physiology Associates, Inc, Fort Myers, Florida
  - Emerald Coast Mood and Memory, PA., Fort Walton Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Mayo Clinic College of Medicine, Jacksonville, Florida
  - Neurology Associates, Maitland, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Pharmax Research Clinic, LLC, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Allied Clinical Trials Inc., Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center, Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - The Roskamp Institute, Inc, Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Johnnie B. Byrd Sr. Alzheimer's Center and Research Institute, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - University of South Florida Suncoast Alzheimer's and Gerontology Center, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, School of Medicine, Atlanta, Georgia
  - Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Medical Research and Health Education Foundation, Inc., Columbus, Georgia
  - Medical Research and Health Education Foundation, Inc, Columbus, Georgia
  - DeKalb Neurology Associates, LLC, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - Maine Medical Partners Neurology, Scarborough, Maine
  - CBH Health, LLC, Rockville, Maryland
  - Brigham and Women's Hospital, Dept. of Neurology, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - ActivMed Practices and Research, Inc., Haverhill, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Donald S. Marks, MD, PC, Plymouth, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Borgess Medical Center/Borgess Research Institute, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Washington University School of Medicine, Saint Lous, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Deaconess Billings Clinical Research Center, Billings, Montana
  - Advanced Neurology Specialists, Great Falls, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - Shore Neurology, PA, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Upstate Clinical Research, LLC, Albany, New York
  - Neurological Associates of Albany, PC, Albany, New York
  - Neuroscience Research Center at Albany Medical Center, Albany, New York
  - Advanced BioBehavioral Sciences, Elmsford, New York
  - Empire Neurology, PC, Latham, New York
  - Neurological Care of Central New York, Liverpool, New York
  - Parker Jewish Institute for Health Care and Rehabilitation, New Hyde Park, New York
  - New York University School of Medicine/Psychiarty, New York, New York
  - Columbia University Medical Center, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center, Monroe Community Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Ohio State University, Dept. of Neurology, Columbus, Ohio
  - Neurology Specialists, Inc., Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Providence Medical Group-Medford Neurology, Medford, Oregon
  - Summit Research Group, LLC, Portland, Oregon
  - Providence Health Service System, AD Center, Brain Institute, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Abington Neurological Associates, Ltd., Abington, Pennsylvania
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Neurology Clinic, P.C., Cordova, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Psychiatric Consultants, PC, Nashville, Tennessee
  - Senior Adults Specialty Research (SASR), Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dept. of Neurology, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - University of Utah, Dept. of Neurology, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - Innovative Clinical Research Center, Alexandria, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Alliance Research Group, LLC, Richmond, Virginia
  - University of Washington Veterans Affairs, Seattle, Washington
  - Pacific Medical Centers, Seattle, Washington
  - Medical College of Wisconsin, Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Landeskrankenhaus- Universitätsklinikum Graz, Graz, Styria, Austria
- Canada (14):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - Medical Arts Health Research Group, Kamloops, British Columbia
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Queens University Memorial Clinics, Kingston, Ontario
  - Parkwood Hospital, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Neurology Research Inc, Toronto, Ontario
  - Toronto Centre for Memory and Aging, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario
  - Neuro Rive-Sud Memory Clinic, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Sir Mortimer B. Davis, Jewish General Hospital, Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Douglas Mental Health University Institute, Verdun, Quebec